CLINICAL TRIAL: NCT01508169
Title: The Effect of Foot Orthoses on the Balance of Elderly Women With Osteoporosis
Brief Title: Foot Orthoses and Elderly Women With Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Ibsen Coimbra, Director of Medical Department of The Faculty of Medical Sciences, State University of Campinas (Unicamp), Brazil, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNICAMP-REUMATO 01
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-02

CONDITIONS: Osteoporosis
Keywords: elderly; balance; insole; foot orthosis; orthotics
MeSH Terms: conditions — Osteoporosis | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foot orthosis (Experimental): Forty-seven women in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas(UNICAMP) who met the inclusion criteria for this study (being female with osteoporosis and aged 60 or above) were assigned, at random, to wear ethyl-vinyl-acetate insoles with medial arch supports and metatarsal pads over a four-week period. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
  Interventions: Device: Foot orthosis (Orthotics Unit of the Clinical Hospital of UNICAMP)
- Control Group (No Intervention): Forty-seven elderly women with osteoporosis (in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas- UNICAMP) were assigned, at random, to enter the control group with no foot intervention. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.

INTERVENTIONS:
Device: Foot orthosis (Orthotics Unit of the Clinical Hospital of UNICAMP) — Custom foot orthoses made of ethylene-vinyl acetate (EVA) with medial arch supports and metatarsal pads (supporting the diaphysis of the second to fourth metatarsals) that were manufactured by the Orthotics and Prostheses Unit of the Clinical Hospital of UNICAMP.
  Other Names: Orthotics Unit of the Clinical Hospital of UNICAMP.
  Arms: Foot orthosis

SUMMARY:
The objective of this study was to determine if foot orthoses are effective in improving balance, pain and disability in elderly women with osteoporosis.

DETAILED DESCRIPTION:
Aging has been associated with balance impairment. The use of foot orthoses has been shown to be a feasible strategy for improving postural control.The objective of this study was to determine if foot orthoses (with metatarsal pad and medial arch support) are effective as an adjuvant treatment to improve balance, foot pain and disability in elderly women with osteoporosis. Another purpose was to verify if social demographic and clinical factors such as age, race, education, marital status, age of menopause, use of drugs related to balance dysfunction, visual or hearing complaints, body mass index, previous fractures and number of falls may influence the results.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of osteoporosis

Exclusion Criteria:

* reduced tactile and thermal foot sensibility
* compromised skin integrity of the lower limbs
* autoimmune rheumatic diseases
* vestibular symptoms
* central nervous system pathologies
* peripheral neuropathy
* use of insoles in the last month
* lower limb prostheses
* previous history of foot surgery
* amputation of the lower limbs
* inability to attend the necessary reevaluations and/or to follow instructions and procedures of the research protocol

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo P Magalhaes, MD, PhD, Study Director — University of Campinas, Brazil; Ibsen B Coimbra, MD,PhD, Study Director — University of Campinas, Brazil; Michael Davitt, Study Director — University of Campinas, Brazil; Cecília M Barbosa, MSc, Principal Investigator — University of Campinas, Brazil; João Francisco Marques-Neto, MD,PhD, Study Director — University of Campinas, Brazil; Manoel B Bértolo, MD,PhD, Study Chair — University of Campinas, Brazil
Locations (1):
- Clinical Hospital of The State University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Meyer PF, Oddsson LI, De Luca CJ. Reduced plantar sensitivity alters postural responses to lateral perturbations of balance. Exp Brain Res. 2004 Aug;157(4):526-36. doi: 10.1007/s00221-004-1868-3. Epub 2004 Mar 17. PMID 15029466
- [Background] Melzer I, Benjuya N, Kaplanski J. Postural stability in the elderly: a comparison between fallers and non-fallers. Age Ageing. 2004 Nov;33(6):602-7. doi: 10.1093/ageing/afh218. PMID 15501837
- [Background] Burke TN, Franca FJ, Meneses SR, Cardoso VI, Pereira RM, Danilevicius CF, Marques AP. Postural control among elderly women with and without osteoporosis: is there a difference? Sao Paulo Med J. 2010 Jul;128(4):219-24. doi: 10.1590/s1516-31802010000400009. PMID 21120434
- [Background] Bernard-Demanze L, Vuillerme N, Ferry M, Berger L. Can tactile plantar stimulation improve postural control of persons with superficial plantar sensory deficit? Aging Clin Exp Res. 2009 Feb;21(1):62-8. doi: 10.1007/BF03324900. PMID 19225271
- [Background] Mulford D, Taggart HM, Nivens A, Payrie C. Arch support use for improving balance and reducing pain in older adults. Appl Nurs Res. 2008 Aug;21(3):153-8. doi: 10.1016/j.apnr.2006.08.006. PMID 18684409
- [Background] Hatton AL, Dixon J, Rome K, Martin D. Standing on textured surfaces: effects on standing balance in healthy older adults. Age Ageing. 2011 May;40(3):363-8. doi: 10.1093/ageing/afr026. Epub 2011 Mar 29. PMID 21450692
- [Background] Palluel E, Nougier V, Olivier I. Do spike insoles enhance postural stability and plantar-surface cutaneous sensitivity in the elderly? Age (Dordr). 2008 Mar;30(1):53-61. doi: 10.1007/s11357-008-9047-2. Epub 2008 Mar 4. PMID 19424873
- [Background] Palluel E, Olivier I, Nougier V. The lasting effects of spike insoles on postural control in the elderly. Behav Neurosci. 2009 Oct;123(5):1141-7. doi: 10.1037/a0017115. PMID 19824780
- [Background] Priplata AA, Niemi JB, Harry JD, Lipsitz LA, Collins JJ. Vibrating insoles and balance control in elderly people. Lancet. 2003 Oct 4;362(9390):1123-4. doi: 10.1016/S0140-6736(03)14470-4. PMID 14550702
- [Background] Wilson ML, Rome K, Hodgson D, Ball P. Effect of textured foot orthotics on static and dynamic postural stability in middle-aged females. Gait Posture. 2008 Jan;27(1):36-42. doi: 10.1016/j.gaitpost.2006.12.006. Epub 2007 Jan 30. PMID 17267222

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2011 to October 2011, patients in treatment in the outpatient clinic of the Rheumatology Division of Unicamp, who met the inclusion criteria for this study (being female with osteoporosis and aged 60 or above) were assessed.
Pre-assignment Details: From the 242 patients considered eligible, 148 were not included due exclusing criteria (compromised skin integrity of the lower limbs, autoimmune rheumatic diseases, vestibular symptoms, central nervous system pathologies, peripheral neuropathy, use of insoles in the last month, previous foot surgery, inability to attend the reevaluations).
Groups:
- Foot Orthosis: Forty-seven women in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas(UNICAMP) who met the inclusion criteria for this study (being female with osteoporosis and aged 60 or above) were assigned, at random, to wear ethyl-vinyl-acetate insoles with medial arch supports and metatarsal pads over a four-week period. Fourty-four subjects completed the protocol.Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
- Control Group: Forty-seven elderly women with osteoporosis (in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas- UNICAMP) were assigned, at random, to enter the control group with no foot intervention. Fourty-five subjects completed the protocol. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
Period: Overall Study
Arm/Group | Foot Orthosis | Control Group
Started | 47 | 47
Completed | 44 | 45
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foot Orthosis | Control Group | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 8 | 12
  >=65 years | 43 | 39 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 72.38 (6.83) | 72.04 (7.14) | 72.38 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 94
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Berg Balance Scale (BBS)
Description: The BBS is a balance assessment test that rates the ability of a subject to maintain balance while performing each of 14 movements required in everyday activities (transferring, standing unsupported, rising from a sitting to a standing position, tandem standing, turning 360° and single-leg standing). Scoring is based on an ordinal 5-point scale from 0 to 4. Total scores ranges from 0 to 56. The smaller value, the worse balance: from 0-20: a whell chair is needed: 20-41: needing walk assistence; 41-56 - independent walking.
Time Frame: 4 weeks
Population: A pilot study (with 14 subjects wearing insoles and 15 controls) was conducted.To identify differences between groups for the variables (Berg, TUG, pain, disability) with a 80% power and a significance level of 5 % the number of 45 subjects in each group was considered satisfactory.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Foot Orthosis: Fourty-seven women in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas(UNICAMP) who met the inclusion criteria for this study (being female with osteoporosis and aged 60 or above) were assigned, at random, to wear ethyl-vinyl-acetate insoles with medial arch supports and metatarsal pads over a four-week period. Fourty-four subjects completed the protocol. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
- Control Group: Forty-seven elderly women with osteoporosis (in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas- UNICAMP) were assigned, at random, to enter the control group with no foot intervention. Fourty-five subjects complited the protocolBalance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
Arm/Group | Foot Orthosis | Control Group
Number analyzed (Participants) | 44 | 45
scores on a scale | 50.68 (4.18) | 43.13 (6.24)

2. Primary Outcome: Timed up and Go Test (TUG)
Description: The TUG test is used to assess the dynamic balance of an individual. It measures the amount of time (recorded in seconds) it takes for the individual to rise from a standard arm chair, walk a distance of 3 meters and return to the initial position resting against the back of the chair.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Foot Orthosis: Forty-seven women in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas(UNICAMP) who met the inclusion criteria for this study (being female with osteoporosis and aged 60 or above) were assigned, at random, to wear ethyl-vinyl-acetate insoles with medial arch supports and metatarsal pads over a four-week period. Fourty-four patients finished the protocol. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
- Control Group: Forty-seven elderly women with osteoporosis (in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas- UNICAMP) were assigned, at random, to enter the control group with no foot intervention. Fourty-five patients finished the protocol. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
Arm/Group | Foot Orthosis | Control Group
Number analyzed (Participants) | 44 | 45
seconds | 11.97 (2.80) | 15.82 (3.23)

3. Secondary Outcome: Numeric Pain Scale
Description: Subjects were asked to rate the pain in their feet on a scale from 0 to 10 (0: no pain, 10: extremely severe pain)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Foot Orthosis | Control Group
Number analyzed (Participants) | 44 | 45
units on a scale | 1.68 (2.46) | 4.20 (3.07)

4. Secondary Outcome: Manchester Foot and Pain Disability Index(MFPDI)
Description: The MFPDI is a test used to assess disability related to foot pain in elderly. It consists of 19 statements prefaced by the phrase "Because of pain in my feet…", organized under three constructs: functional limitation (10 items), pain intensity (five items), and personal appearance (two items). For each statement, there are three possible answers: "none of the time" (score = 0), "some days" (score = 1), and "most days/every day" (score = 2). The final score is the sum of all the items and ranges from 0 to 38. The higher score, the greater disability.
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Foot Orthosis: Forty-seven women in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas(UNICAMP) who met the inclusion criteria for this study (being female with osteoporosis and aged 60 or above) were assigned, at random, to wear ethyl-vinyl-acetate insoles with medial arch supports and metatarsal pads over a four-week period. Fourty-four patients completed the protocol. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
- Control Group: Forty-seven elderly women with osteoporosis (in treatment in the outpatient clinic of the Rheumatology Division of State University of Campinas- UNICAMP) were assigned, at random, to enter the control group with no foot intervention. Fourty-five patients completed the protocol. Balance, using the Berg Balance Scale (BBS) and the Timed Up and Go (TUG) indexes; pain, using a numeric pain scale (NPS); and disability of the feet, using the Manchester Foot Pain and Disability Index (MFPDI), were assessed at baseline and after four weeks.
Arm/Group | Foot Orthosis | Control Group
Number analyzed (Participants) | 44 | 45
scores on a scale | 11.48 (5.56) | 22.64 (9.20)

ADVERSE EVENTS:
Time Frame: The subjects from the foot orthoses group were asked to note and report the occurrence of any adverse effects during a four-week period.
Arm/Group | Foot Orthosis | Control Group
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/0
Other Adverse Events (participants affected / at risk) | 6/47 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foot Orthosis (N=47) | Control Group (N=0)
foot discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
feet heat (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
tightness of footwear (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No